CLINICAL TRIAL: NCT01949896
Title: Impact of Feeding on Pro-Inflammatory Cytokine Response in Neonates Receiving a RBC Transfusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is being closed due to insufficient patient population for enrollment.
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Andrew Ellefson, MD / Neonatal Fellow, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DDD602270
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Transfusions
Keywords: Pro inflammatory cytokine; Necrotizing enterocolitis; Packed red blood cell transfusion
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: NPO (Other): Infants in this group will be made NPO approximately 4 hours prior to receiving a blood transfusion and will remain NPO until approximately 24 hours after the blood transfusion.
  Pro-inflammatory cytokine response will be monitored at 3 times points.
  Interventions: Other: NPO
- Control: Continue feedings (Other): Infants in this group will be allowed to continue feedings during the transfusion at the discretion of the medical team.
  Pro-inflammatory cytokine response will be monitored at 3 times points.
  Interventions: Other: Control group: continue feedings

INTERVENTIONS:
Other: NPO — Infants in this group will be made NPO for a period of time surrounding the packed red blood cell transfusion.
  Arms: Intervention: NPO
Other: Control group: continue feedings — Feedings will be continued in this group.
  Arms: Control: Continue feedings

SUMMARY:
Prior to a non-urgent blood transfusion, subjects will be randomized to either stopping feeds or continuing feeds. The intervention group will be the placement of a subject in the NPO group. Subjects in the intervention group will have their feedings stopped for a total of 24 hours around the time of the PRBC transfusion. These infants will be given intravenous nutrition during the period of time that they will not be fed. During the transfusion, both groups of subjects will have serum cytokine levels obtained at 3 time intervals- 1) 4 hours pre-transfusion, 2) 2-4 hours post-transfusion, and 3) 20-24 hours post-transfusion.

DETAILED DESCRIPTION:
Recently many publications have indicated a potential temporal association between packed red blood cell (PRBC) transfusion and the development of NEC in neonates. Although, to date, there is no conclusive evidence indicating a causal role of PRBC transfusion on the development of NEC. Given the growing body of data that support the association of PRBC transfusions and NEC, a common clinical dilemma arises with regard to feeding infants during a blood transfusion. Additionally, it is thought that increased immunomodulation may be exacerbated by any other pro-inflammatory process or insult; thereby leading to a rapidly increasing cascade of pro-inflammatory cytokines which may ultimately lead to gut inflammation and NEC.

Prior to a non-urgent PRBC transfusion, subjects will be randomized to either the NPO group or fed group of patients. The intervention will be the placement of a subject in the NPO group. Subjects will be made NPO for a total of 24 hours around the time of the PRBC transfusion. During the transfusion, both groups of subjects will have serum cytokine levels obtained at 3 time intervals- 1) 4 hours pre-transfusion, 2) 2-4 hours post-transfusion, and 3) 20-24 hours post-transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Infants born < 31 weeks gestational age
* Between 3 and 7 days old at time of consent

Exclusion Criteria:

* Infants with multiple congenital anomalies
* Infant with suspected/confirmed genetic anomalies
* Infant with suspected/confirmed congenital immune deficiencies

Ages: 3 Days to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pro-inflammatory cytokine response | 24 hours
  Evaluate the pro-inflammatory cytokine response in both fed and NPO infants during a transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ellefson, MD, Principal Investigator — Christiana Care Health Services; David A Paul, MD, Study Director — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States